CLINICAL TRIAL: NCT02420678
Title: Validation of Questionnaire Module for Quality of Life and Analysis of Its Association With Clinical Outcomes; a Cohort Study in Patients With Hepatocellular Carcinoma
Brief Title: Quality of Life in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ju Hyun Shim, Assistant Profesor, Asan Medical Center
Other Study IDs: AMC 2015-0229
Record Dates: First submitted 2015-03-26; First posted 2015-04-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the second leading cause of cancer-related mortality worldwide. Despite the recent advances in the treatment of HCC, the prognosis of HCC is still poor even after curative treatment.

Performance status has shown to be associated with long-term survival and prognosis in patients with HCC, and it is one of the important factors in the Barcelona Clinic Liver Cancer (BCLC) staging system. Recently, the researches on health-related quality of life (HRQL) of cancer patients have been progressed. The most widely used surveys to assess HRQL of cancer patients are Functional Assessment of Cancer Therapy-Generic (FACT-G) and European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30. Since those two are mainly about cancers in general, HCC specific surveys were developed.

The FACT-Hep questionnaire has 45-items specifically focusing on patients with hepatobiliary cancers. EORTC QLQ-hepatocellular carcinoma 18 (HCC 18) is an 18-item questionnaire designed to be used along with the EORTC QLQ-C30 for patients with HCC. An 18-item National Comprehensive Cancer Network (NCCN)-FACT Hepatobiliary-Pancreatic Symptom Index (NFHSI-18) is a specific questionnaire for advanced hepatobiliary and pancreatic cancers. However, there is no consensus whether it would be appropriate to adopt HRQL as a prognostic variable in HCC staging system. Moreover, there is limited information available about the impact of patients' HRQL on long-term outcome in patients with HCC.

Thus, in this study, the researchers will investigate whether HRQL can be an important factor in HCC staging system by testing the reliability and clinical validity of FACT-Hep, EORTC QLQ-HCC18, and NFHSI-18. Second, the investigators will evaluate the relation of HRQL with treatment efficacy, recurrence and survival outcome. Lastly, the investigators will suggest the suitable questionnaire module for patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of HCC
* Ability to speak, read, and write Korean
* Patient is able and willing to give informed consent

Exclusion Criteria:

* Evidence of cognitive impairment or psychiatric disturbance
* Other concurrent malignancy
* Patients involved in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted hepatocellular carcinoma (HCC) patients will be screened to determine study eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical validity of FACT-Hep, EORTC QLQ-HCC18 and NFHSI-18 | Baseline
  The FACT-Hep questionnaire consists of 18-item Hepatobiliary Subscales and 27-item FACT-G, which contains physical (7 items), social (7 items), emotional (6 items), and functional scales (7 items). Hepatobiliary Subscale is scored 0-72, FACT-G is scored 0-108, and FACT-Hep is scored 0-180. EORTC QLQ-HCC 18 is an 18-item questionnaire designed to be used along with the 30-item EORTC QLQ-C30. EORTC QLQ-HCC 18 questionnaire includes 8 symptom scales such as fatigue, jaundice, nutrition, pain, fever, abdominal swelling, sexual interest, and body image. Each item is scored 0-100 according to the EORTC guidelines. NFHSI-18 consists of 18-item scales, and each item is scored 0-4, yielding a total between 0 and 72. The investigators will test the validity by using the correlation and comparison of all of the questionnaire scores at baseline.
Reliability of FACT-Hep, EORTC QLQ-HCC18 and NFHSI-18 | Baseline and at least 6 hours later
  Patients will complete the questionnaires at baseline and then will respond to the follow-up surveys at least 6 hours later the first assessment. The investigators will examine reliability by assessing test-retest reliability of each survey after measuring the scores of questionnaires at two assessment points.

SECONDARY OUTCOMES:
Recurrence rates | upto 3 years
Death rates | upto 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ju Hyun Shim, MD, PhD, Principal Investigator — Gastroenterology, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea